CLINICAL TRIAL: NCT04558723
Title: Randomized Controlled, Multi-centre Trial of Cardiac Magnetic Resonance Guidance of Implantable Cardioverter Defibrillator Implantation in Non-ischemic Dilated Cardiomyopathy
Brief Title: Cardiac Magnetic Resonance Guidance of Implantable Cardioverter Defibrillator Implantation in Non-ischemic Dilated Cardiomyopathy
Acronym: CMR-ICD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. med. Ingo Eitel (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Ingo Eitel, Director, University of Luebeck
Organization: University of Luebeck (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-275; CMR-ICD-DZHK23 (Other: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK))
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Non-ischemic Dilated Cardiomyopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICD group (Experimental): Patients receiving OMT and ICD or cardiac resynchronization therapy with a defibrillator (CRT-D) if indicated.
  Interventions: Other: ICD/CRT-D implantation
- Optimal HF care group (No Intervention): Patients receiving OMT and CRT pacemaker (CRT-P) implantation without a defibrillator if indicated. Patients without CRT indication will receive an ICM for detection of malignant VAs.

INTERVENTIONS:
Other: ICD/CRT-D implantation — ICD/CRT-D implantation (if indicated)
  Arms: ICD group

SUMMARY:
Patients with diagnostic CMR images for assessment of LGE/fibrosis and evidence/presence of non-ischaemic myocardial fibrosis/scar will be randomized to the following treatment groups in a 1:1 ratio: ICD group or Optimal HF care group.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the hypothesis that implantable cardioverter defibrillator (ICD) therapy would decrease the risk of death from any cause in comparison to optimal heart failure (HF) care without ICD insertion in patients with NIDCM, left ventricular ejection fraction (LVEF) ≤35% and presence of myocardial fibrosis on cardiac magnetic resonance (CMR) imaging.

ELIGIBILITY:
Inclusion Criteria:

* NIDCM (idiopathic or familial)*
* LVEF ≤35% and presence of fibrosis on CMR
* Diagnostic CMR scan
* Age ≥18 years
* Written informed consent
* Ability to give informed consent

Exclusion Criteria:

* ICM [previous myocardial infarction, previous percutaneous coronary intervention]
* Other cardiomyopathies (hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, infiltrative cardiomyopathies [e.g. cardiac amyloidosis, cardiac sarcoidosis, hemochromatosis and iron overload cardiomyopathy], left ventricular non-compaction cardiomyopathy, reversible cardiomyopathies [Takotsubo syndrrome, peripartum cardiomyopathy, chemotherapy induced cardiomyopathy].
* Myocarditis
* Contraindication for CMR at study entry (including severe claustrophobia, pacemaker or ICD, metallic cerebral or intracranial implants, known allergy to gadolinium)
* Severe renal insufficiency (creatinine clearance <30 mL/min)
* Current pacemaker or defibrillator in situ
* Current indication for device therapy (e.g. secondary prophylaxis after aborted SCD)
* Renal impairment defined as an eGFR <30 milliliters
* Age <18 years
* Patients presenting with pregnancy
* Patients without informed consent
* Participation in another randomized trial
* Life expectancy <2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Death from any cause | Day 0
  Death from any causes during follow-up - after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Ingo Eitel, Prof. Dr., Principal Investigator — Medical Clinic II - University Heart Center Lübeck
Locations (1):
- Universität zu Lübeck, Lübeck, Schleswig-Holstein, Germany